CLINICAL TRIAL: NCT05403359
Title: Optimal Dosing and Timing of Corticosteroids in Hospitalized Patients With COVID-19.
Brief Title: StEroids in hospitaLized patiEnts With Covid-19 in The Netherlands.
Acronym: SELECT
Status: Completed | Type: Observational
Sponsor: Henrik Endeman (Other)
Collaborators: Amsterdam UMC (Other); OLVG (Network); Isala (Other); St. Antonius Hospital (Other); Academisch Ziekenhuis Groningen (Other); Amphia Hospital (Other); Maasstad Hospital (Other)
Responsible Party: Sponsor-Investigator, Henrik Endeman, Principal investigator, Erasmus Medical Center
Organization: Erasmus Medical Center (Other)
Other Study IDs: 10430102110010
Record Dates: First submitted 2022-06-01; First posted 2022-06-03 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Steroids

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Ward (e.g., pulmonology ward, COVID-unit, etc.),: * WP1A: Patients with WHO clinical progression scale class 4-5 (i.e., no oxygen therapy) admitted to the ward with laboratory-confirmed COVID-19.
  * WP1B: Adult patients admitted to the ward with laboratory-confirmed COVID-19 and on at least oxygen therapy.
  Interventions: Drug: Steroids
- Intensive Care Unit: Adult patients (≥18 years) admitted to the ICU with laboratory-confirmed COVID-19 and acute respiratory distress syndrome (ARDS) according to the Berlin definition criteria (i.e., receiving invasive mechanical ventilation).
  Interventions: Drug: Steroids

INTERVENTIONS:
Drug: Steroids — Description of the intervention in each of the work packages:
  * WP1A admission: Steroid dose >6mg/day dexamethasone equivalent will be compared to control (steroid = 6mg/day dexamethasone or equivalent steroid).
  * WP1B late: After 10 days of dexamethasone therapy patients are stratified in high-dose steroids (> 6 mg dexamethasone or equivalent steroid) or no steroids up to day 28.
  * WP2 ICU admission: High-dose steroids (dexamethasone >6 mg daily or equivalent corticosteroids) compared to dexamethasone 6 mg up to 72 hours after admission
  * WP3 ICU late: After dexamethasone 6 mg for 10 days patients are stratified in high-dose steroids (dexamethasone >6 mg daily or equivalent corticosteroids) or no steroids up to day 28.

SUMMARY:
Rationale: In patients with COVID-19 admitted to the hospital, large heterogeneity exists in patients, timing and dosing of steroid therapy. It is unclear how to treat patients who fail dexamethasone therapy. High-dose steroids are prescribed mainly in patients with the most severe disease, which may be too late given the potential escalation of pathophysiological pathways in these patients.

Objectives: The main objective is to determine the most optimal form, timing and dosing of steroid therapy to reduce the morbidity and mortality of patients admitted to the hospital for COVID-19. This objective will be addressed in 4 work packages (WP):

* WP-1A-ward admission: What is the effect of higher dose steroids upon hospital admission on clinical deterioration and what would be the optimal timing of increasing steroid dosage?
* WP1B-ward late: Do high-dose steroids, compared to no steroids, improve outcomes in dexamethasone-unresponsive COVID-19 patients on the ward after dexamethasone 6 mg/day for 10 days?
* WP2-ICU admission: Do high-dose steroids, compared to 6 mg/day dexamethasone or its equivalent, improve outcomes in patients admitted to the ICU with moderate/severe C-ARDS?
* WP3-ICU late: Do high-dose steroids, compared to no steroids, improve outcomes in ICU patients with moderate/severe C-ARDS after dexamethasone 6 mg/day for 10 days?
* WP4-biobank: Can biomarkers help predict outcomes after (high dosed) steroid therapy? Study design: Retrospective observational multicenter study in the Netherlands.

Study population: Adult patients (≥ 18 years) hospitalized with COVID-19 will be included, more specifically:

Intervention (if applicable): Not applicable (retrospective study design).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: Given the retrospective nature of the study, no burden, risks or benefits for the patient are associated with participation. The target population of this study is specific to hospitalized patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria:

To be eligible for inclusion in any of the work packages, an individual must meet all of the following general inclusion criteria:

1. Adult (i.e., ≥18 years)
2. Hospitalized (i.e., admitted to the hospital)
3. Laboratory-confirmed COVID-19 diagnosis (i.e., based on polymerase chain reaction-(PCR) test)

WP1A- ward early:

(1) Patients who present with WHO clinical progression scale class 4-5 (no oxygen therapy, Figure 5) when admitted to the ward with COVID-19.

WP1B-ward late:

1. Admitted to the ward (e.g., pulmonology ward, COVID-unit, etc.), excluding step-down units.
2. In need of non-invasive oxygen therapy during hospital stay, including:

   * Conventional oxygen therapy (COT) 1-5 L/min
   * Conventional oxygen therapy (COT) 6-12 L/min
   * Non-rebreather mask 12-15 L/min
   * High-flow nasal cannula 16-60 L/min
   * Non-invasive continuous positive airway pressure (CPAP)
   * Non-invasive bilevel positive airway pressure (BiPAP)

WP2-ICU admission/ WP3-ICU late:

1. Admitted to the ICU>48 hours.*
2. Invasive mechanical ventilation during ICU stay (intubation with endotracheal tube or tracheostomy) or extracorporeal membrane oxygenation (ECMO).
3. ARDS according to the Berlin criteria

WP4-biobank:

The study population consists of patient subsets admitted to the ICU described in WP2 and WP3.

Exclusion Criteria:

General exclusion criteria:

* Mortality within 48 hours.*
* Opt-out (objection to participate)

Criteria indicated with an asterisk (*) may or may not be applied, depending on data availability. These criteria will be instated if they result in excessive variation of the outcome or exposure, or result in difficulty in generalizing to the target population.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) hospitalized with laboratory-confirmed COVID-19.The (hospitalized) study population is expected to consist mainly of older, male, obese patients who suffer from comorbidities, like hypertension, diabetes mellitus. Around 40% of these patients require invasive mechanical ventilation. The investigators will include patients from all SARS-CoV-2 epidemic waves (including the first wave).
Sampling Method: Probability Sample
Enrollment: 2465 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2023-12-01 (Actual)

PRIMARY OUTCOMES:
28-day survival (WP2-3) | Day 28
  Alive at day 28 yes/no
28-day need of invasive mechanical ventilation (WP2-3) | Day 28
  Need for mechanical ventilation at day 28 yes/no
Need for WHO severity 6-9 (WP1) | From date of hospital admission up to date of hospital discharge, assessed up to 12 months
  WHO clinical progression scale class 6: high flow nasal cannula WHO class 7-9: invasive ventilation
Hospital mortality in patients who receive HFNC or invasive mechanical ventilation due to restrictions in care (WP1) | From date of hospital admission up to date of hospital discharge, assessed up to 12 months
  Restrictions in care (either on medical grounds or by advance directive of the patient)

SECONDARY OUTCOMES:
ICU mortality | During ICU stay
  Death at ICU including date
Hospital mortality | From date of hospital admission up to date of hospital discharge, assessed up to 12 months
  In-hospital death including date
Hospital length of stay | From date of hospital admission up to date of hospital discharge, assessed up to 12 months
  The number of days from the date of hospital admission to date of hospital discharge or death
ICU length of stay | During ICU stay
  The number of days from the date of ICU admission to date of ICU discharge or death
Mechanical ventilation duration | During ICU stay
  Total duration of mechanical ventilation in days
Ventilator free days and alive | Day 28
  Number of ventilator free days at day 28
Rate of respiratory and inflammatory complications during hospital stay | From date of hospital admission up to date of hospital discharge, assessed up to 12 months
  Aspergillus, Herpes simplex virus (HSV),Cytomegalovirus (CMV), Ventilator-associated pneumonia (VAP), Catheter-related bloodstream infection (CRBSI)
Rate of general systemic complications during hospital stay | From date of hospital admission up to date of hospital discharge, assessed up to 12 months
  Myocardial infarction, deep venous thrombosis, pulmonary embolus, hyperglycemia, hypoglycemia, acute kidney injury, delirium, sepsis

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, Rotterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available through a secure data transfer system and appropriate data transfer agreement. (The data set contains personal data.)
Supporting Information: Study Protocol
Access Criteria: Reasonable requests via email (including a protocol describing the research question and data needed) are considered.

REFERENCES:
- [Derived] Daenen K, Rizopoulos D, Dalm VASH, Huijben JA, Stoof SCM, Nagtzaam NMA, Dik WA, Swagemakers SMA, van der Spek PJ, Tong-Minh K, Mersha DGA, Khyali J, Juffermans NP, Gommers D, van Gorp ECM, Bos LDJ, Endeman H. Increasing inflammatory biomarkers are associated with mortality in critically ill COVID-19 patients despite anti-inflammatory treatment. Clin Exp Med. 2025 Nov 11;25(1):361. doi: 10.1007/s10238-025-01904-8. PMID 41217548
- [Derived] Daenen K, Huijben JA, Boyd A, Bos LDJ, Stoof SCM, van Willigen H, Gommers DAMPJ, Moeniralam HS, den Uil CA, Juffermans NP, Kant M, Valkenburg AJ, Pillay J, van Meenen DMP, Paulus F, Schultz MJ, Dalm VASH, van Gorp ECM, Schinkel J, Endeman H; PRoVENT- and PRoAcT-COVID Collaborative Group. Optimal Dosing and Timing of High-Dose Corticosteroid Therapy in Hospitalized Patients With COVID-19: Study Protocol for a Retrospective Observational Multicenter Study (SELECT). JMIR Res Protoc. 2023 Jun 2;12:e48183. doi: 10.2196/48183. PMID 37266993